CLINICAL TRIAL: NCT07117643
Title: Influence of Remote Ischemic Preconditioning Reperfusion/Reocclusion Training and Physical Exercises on the Inflammatory, Angiogenic, Neurotrophic and Anti-tumor Potential of Human Serum in Vivio/in Vitro Studies - Role of Vitamin d and Iron Metabolism
Brief Title: Ischemic Preconditioning - Perspectives of Use Vivio/in Vitro Studies
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Gdansk University of Physical Education and Sport (Other)
Collaborators: Medical University of Gdansk (Other); Kazimierz Wielki University (Other); Università Politecnica delle Marche (Other); Charles University, Czech Republic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: AWFiS/2025_7_JM; 2/16/12/2024 (Other: University of Physical Education and Sport (GUPES))
Record Dates: First submitted 2025-07-16; First posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-07

CONDITIONS: Sport Medicine; Sport; Physiological Adaptations; Sport Performance; Remote Ischemic Preconditioning; Ischemic Preconditioning
Keywords: inflammation; remote ischemic preconditioning; hepcidin; Iron; erytropheron; RIPC; IPC
MeSH Terms: conditions — Inflammation | interventions — Ischemic Preconditioning; Reperfusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 1-time SHAM intervention (Sham Comparator): 1 time SHAM intervention
  Interventions: Other: Ischemic Preconditioning
- 10-time SHAM intervention (Sham Comparator): 10-time SHAM intervention
  Interventions: Other: Ischemic Preconditioning
- 1-time RIPC intervention (Experimental): 1-time RIPC intervention on anaerobic/aerobic performance
  Interventions: Other: Ischemic Preconditioning
- 10-time RIPC intervention (Experimental): 10-time RIPC intervention on anaerobic/aerobic performance
  Interventions: Other: Ischemic Preconditioning

INTERVENTIONS:
Other: Ischemic Preconditioning — The ischemic procedure will be carried out before the start of the WanT and eccentric exercises procedures and muscle damage in accordance with the detailed description of the RIPC procedure. Four-fold filling of the flotation flange will be performed by 5 minutes to the value of 200 mm Hg with 5 minutes' rest interval near the attachment of the initial straight thigh muscle. All performed procedures will be carried out under the Doppler USG control to perform full arterial blood flow restriction.
  The whole research will be carried out in the Laboratory in morning hours. Each participant will be in a hydrated state and before the first meal.
  Other Names: IPC; RIPC; REPERFUSION/REOCCLUSION TRAINING

SUMMARY:
Both in sports and medicine, methods that can significantly contribute to improving the ability of tissues to perform their functions are constantly being searched. One of those methods that is increasingly used also in sports is remote ischemic preconditioning (RIPC). Mostly, this procedure involves repeated brief cycles of limb ischemia/reperfusion. This method is often referred as ischemic blood reperfusion and helps to increase the tolerance of treated tissues to the occurrence of possible ischemic episodes in the future. Numerous studies have shown that RIPC induces changes that lead to increased resistance to hypoxia and other stressors in organs (brain, heart, liver). In addition, it has been proven that induction of arterial occlusion in the area of selected limbs before performing physical exercises can affect the improvement of their function, and thus can translate into sports results. In addition, an adaptation of such fibres to damage is mostly associated with the secretion of many factors that influence body function. That's why we conclude that it may affect protein kinases (such like c-Jun N-terminal kinases (JNKs) or serine-threonine kinase = protein kinase B (AKTs)) whose main role is regulation of the activity of a wide spectrum of substrates, influencing cells proliferation, apoptosis, responses to cellular stress and inflammatory process in normal and cancer cells. Concluding that presented kinases activity is associated with cells differentiation and RIPC and physical activity may affect them and the inflammation process that may lead to cytotoxic activity against cancer cells (especially if the effects are combined together). The beneficial increase of anti-tumour activity of the blood serum against pathological isolated tumour cells of prostate cancer (cell lines - LNCaP and PC- 3) was confirmed in our pilot studies. We observed an increase in the anti-cancer properties of serum taken from people that attended RIPC training and performed physical activity. However, the exact mechanism and associated changes in the proteome of blood serum people attending in the RIPC training have not yet been determined. This knowledge would allow us to determine the exact mechanisms of the reperfusion/reocclusion training on the human body and its beneficial activity. Considering that the skeletal muscle is an organ capable of synthesis and release of a number of proteins, cytokines and low molecular weight compounds, especially during physical activity, it should be assumed that intermittent muscle ischemic episodes will lead to increased release of factors that will increase the resistance of muscles and other tissues to stress. At the same time, it was noticed that under conditions of muscular stress induced changes in iron metabolism occur. The binding of free iron through the ferritin protein at the cell level leads to its greater resistance to stressors. In the prism of the above considerations, the results of our preliminary studies showing that the upper limb RIPC procedures cause changes in iron metabolism in white blood cells and may suggest that the procedure of RIPC leads to changes that allow storing iron in a safe form in as ferritin. At the same time, with the increasing interest in iron metabolism, the role and function of amyloid precursor protein (APP) and hepcidin are increasing. It has been proven that APP is a protein that works with ferroportin, thus taking part in iron export from a cell. Moreover, it has been shown that the post-translational modification of APP leads to the formation of amyloid α (determines positive changes) and amyloid β (negative changes). Because there are some indications that sAPPα may be modified by iron changes and associated with cfDNA changes, which substantially increase during i.e. tissue damage, we would like to explore those correlations more deeply. The same decrease in the APP protein level will lead to the inhibition of iron export from the cell and an increase of its concentration in the cell. The nature of such changes in iron metabolism should be considered as adaptive to the ischemic stress on which muscle is exposed during the RIPC procedure. The increase in ferritin in the cell leads to a decrease in the concentration of free iron and thus a reduction in iron-dependent ROS formation. This project will have an impact on the development of the current state of knowledge of the mechanisms of biochemical response to the specific tissue-affecting method in form of remote ischemic preconditioning and will allow determining the role of sAPPα and Cathepsin C and other trophic factors and changes in iron metabolism in this process, taking into account the role of hepcidin and vitamin D. Moreover, the present project may contribute to the determination of the role of presented procedures on cells proliferation, as an example of anti-tumour proprieties, and changes of human serum proteomes.

DETAILED DESCRIPTION:
Both in sport and medicine, constantly new methods are being search that can significantly improve the ability of tissues to perform their functions. One of such methods, increasingly used also in sport an physical activity is the Remot Ischemic Preconditioning (RIPC). In most cases, this procedure involves repeated brief cycles of limb ischemia and reperfusion. And often is being said that it helps to increase the tolerance of treated tissues to the occurrence of possible ischemic episodes in the future. Numerous studies have shown that RIPC induces changes that lead to increased resistance to hypoxia and many other tissue stressors in numerus organs, such as brain, heart, liver, kidneys etc.

In addition, in case of skeletal muscles, it has been proven that induction of arterial occlusion in the part of selected limbs before performing physical exercises can affect its activity by causing the improvement of its function and performance, and thus can result in to a sports scores (results). In addition, a greater resistance of such fibers to damage induced by eccentric contractions was observed. The mechanism of this method, however, is not fully understood, and its character can be very complex and effects tissue on many stages of its activity.

On the other hand considering that the skeletal muscle is an endocrine organ capable to synthesis and release a number of proteins, cytokines and low molecular weight compounds, especially during physical activity, it should be assumed that that intermittent muscle ischemic episodes will lead to increased release of factors that will increase the resistance of muscles and other tissues to stress.

In addition, adaptation of such fibers i mostly associated with the secretion of many factors that influence whole body function.

One of such substances are protein kinases. They are responsible for regulation of many biological processes, as well as a molecularly targeted anti-cancer therapy due to the increased level it's activity in many cancers. These enzymes carry out the phosphorylation reaction of a specific molecules. Phosphorylation usually changes the conformation of the protein molecules and, consequently, changes its activity, and ability to bind to other proteins, or the movement of the molecule within the cell. Most research indicates that they play a key role in many fundamental cellular processes such as the cell cycle, cell division, differentiation and apoptosis. Deregulation of kinase activity as a result of chromosomal mutations, rearrangements and / or gene amplification is observed in many types of cancer cells. Therefore, such procedures like RIPC or intensive physical activity that could affects it's activity may be specific inhibitors of these enzymes, fulfilling the idea of molecularly targeted therapy. Therefore, we conclude that it may affect some specific protein kinases (such like c-Jun N-terminal kinases (JNKs) or serine-threonine kinase = protein kinase B (AKTs)), and may be associated with cancer cells life, especially if the effect is combined together (RIPC + physical activity). Therefore, in our pilot studies, we assessed the effect of the 10 days RIPC procedure on the anti-tumor potential of human serum in relation to the prostate tumor line LNCaP. We observed statistical significance increase of human serum antitumor potential which may be connected to the effect on protein kinase pathways. However, this requires further confirmation and analyzes of a larger population of people subjected to the RIPC procedure and physical activity. From this research it's seems advisable to assess whether the ischemic procedures affects antitumor properties of human serum by itself or is it connected to the impact of other factors such like physical activity.

At the same time, it was noticed that under conditions of muscular stress induced changes in iron metabolism occur. Iron is a metal that is necessary for almost all cell processes and, on the other hand, it can be very toxic - stimulating the formation of reactive oxygen species (RFT). Binding of free iron through the ferritin protein at the cell level leads to its greater resistance to stressors. In the prism of the above considerations, the results of our preliminary studies showing that the upper limb RIPC procedures used in case of young men causes changes in iron metabolism in white blood cells. We observed that RIPC increase ferritin genes and protein level in WBC. Increase in ferritin H protein level was shown to reduce labile iron pool and iron-dependent ROS formation. These data suggest that the procedure of remote ischemic preconditioning induced adaptive changes is associated with changes in iron metabolism.

At the same time, with the increasing interest about iron metabolism the role and function of amyloid precursor protein (APP) and hepcidin is increasing. It has been proven that APP is a protein that works with ferroportin, thus taking part in iron export from a cell. Moreover, it has been shown that the post-translational modification of APP leads to the formation of amyloid α (determines positive changes) and amyloid β (negative changes). Numerous beneficial effects of the action of amyloid α in the human body has been shown (increase in insulin sensitivity, neurotrophic effect, stimulation of synaptogenesis) tend to seek methods for inducing its secretion. In addition, an increase in sAPPα concentration will be associated with a decrease in the membrane form of APP.

The same decrease in the APP protein level will lead to the inhibition of iron export from the cell and increase of its concentration in the cell. The nature of such changes in iron metabolism should be considered as a adaptive to the ischemic stress on which muscle is exposed during the RIPC procedure. The increase in ferritin in the cell leads to a decrease in the concentration of free iron and thus a reduction in iron dependent ROS formation. In addition, the reduction of iron export from the cell will lead to a decrease in its concentration in the extracellular fluid and blood, which may also increase tolerance to stress.

Hepcidin, induces a suppressive effect on ferroportin, limiting the absorption of iron from the gastrointestinal tract as well as its release from intra-human body system resources, including liver and macrophages. The concentration of hepcidin in the blood increases during inflammation. It seems that the main goal of this increase is to limit the availability of iron, which in the free form has a pro-inflammatory effect and can stimulate the development of pathogens.

It has been shown so far that staying under hypoxia conditions leads to a decrease in the concentration of hepcidin, which is aimed at ensuring adequate supply of iron to the increasing erythropoiesis. These changes are associated with increase in EPO which will stimulate erythroblasts to produced ERFE and it will inhibit hepcidin biosynthesis. In turn, the barrack is data whether the RIPC procedure will induce substitution in hepcidin, ERFE and EPO concentration. In turn, there is no data if the RIPC procedure will induce substitution at the hepcidin concentration. Similar there is no data how in this situation postconditioning procedure can affect hepcidin concentration and the formation of amyloid α.

Vitamin D plays a crucial role in the regulation of multiple physiological processes. Its activity is mainly ascribed to the active form, 1,25(OH)2D3, which acts via a specific vitamin D receptor (VDR). VDR is a transcriptional factor that regulates the expression of approximately 1000 genes. VDR is present in almost all human tissues (Wang et all. 2012). Vitamin D is produced in the skin in response to ultraviolet (sunlight) exposure. Subsequently, it is hydroxylated at positions 25 and 1 to gain full hormonal activity.

On the other hand, 25-OH vitamin D [25(OH)D3] is a good marker of vitamin D status. The kidney, brain, bone, skin, prostate, and white blood cells can convert 25(OH)D3 to its active form [1,25(OH)2D3]. It can be anticipated that low serum levels of 25(OH)D3 will limit the synthesis of the active form in all these tissues. Serum 25(OH)D3 levels are mainly determined by the exposure to sunlight and vitamin D supplementation. In addition, higher fat tissue content is associated with lower serum 25(OH)D3 levels, possibly because of its ability to store vitamin D. On the other hand, higher physical activity is associated with better vitamin D status, even though many athletes are vitamin D-deficient. Collectively, the above observations indicate that vitamin D metabolites have important biological functions, which are far from being completely understood. On the other hand, there was still lack of knowledge about muscles activity and Vitamin D concentration. The key discovery that pointed to a role for muscle in maintaining vitamin D status came from studying the properties of muscle cells in vitro. The cell membrane was found to contain the proteins megalin and cubilin. These proteins, like those in the renal tubule cells and in hepatic stellate cells, transport DBP from the extracellular fluid into the cell cytoplasm.

The vitamin D binding protein has two specific, high-affinity binding sites. One is for vitamin D and its metabolites with the highest affinity being for 25(OH)D. The other binding site is specific for filamentous actin. A commonly held theory postulates that the actin-binding site of DBP functions to bind actin if released into blood from damaged cells and, thus, protects against intravascular coagulation. Yet it has been known for over 30 years that DBP becomes bound to actin in skeletal muscle. Some of the internalized DBP could be bound to actin in actomyosin, via its specific actin-binding site, but much of the remainder is bound to actin dispersed throughout the cytoplasm.

Since then, many more studies have been conducted, and the mechanisms of vitamin D have become increasingly clear. Nevertheless, how vitamin D affects exercise has not been thoroughly discussed. Currently, we know that muscle performance lowers vitamin D deficiency in exercisers. These results indirectly demonstrate that vitamin D potentially affects exercise performance; however, whether vitamin D reduces exercise-induced damage or the oxidative stress caused by exercise requires confirmation.

Therefore, it is crucial to study the effects of exercise on vitamin D metabolism. Exercise stimulates the release of several hundreds of proteins (myokines) into the circulation from the skeletal muscle, while also stimulating the liberation of bioactive proteins (exerkines) from other tissues. An example of such exerkine is fibroblast growth factor 23, whose concentration increases after exercise. This exerkine is responsible for the regulation of plasma phosphate levels and modifies vitamin D metabolism by inhibiting the formation of 1,25(OH)2D3 (Shimada et all., 2004). Therefore, it seems important to assess the effect of vitamin D concentration on the level of post-exercise muscle damage and the relationship between its concentration and iron concentration and the induced inflammatory process that's occurs after physical activity.

Recent years brought the era of cell-free DNA (cfDNA) as a potential biomarker of the level of injury, which is gaining interest in many various biomedical disciplines, including the field of exercise physiology. There are more and more studies looking for the role of cDNA as a potential hallmark of the overtraining syndrome in: resistance training, marathon run, continuous treadmill running, incremental exercise, rowing exercise, strength training.

Besides cfDNA might be related to, or trigger adaptations of immune function induced by strenuous exercise. Publication from 2017 revealed an increase cfDNA level even during aerobic running below the lactate steady state depending on intensity and duration. It was observed that cfDNA concentrations peaked immediately after acute exercise and about 1h post-exercise returned to baseline levels. Furthermore, typical markers of skeletal muscle damage (C-reactive protein, uric acid, creatine kinase, myoglobin) display delayed kinetics compared with the cfDNA peak response. All of that underlines the potential of cfDNA as a biomarker for exercise load in both -the aerobic and the anaerobic state. However there was not much effort put into finding the correlations between cfDNA and iron state and exercises induced inflammation process.

This project will have an impact on the development of the current state of knowledge of the mechanisms of biochemical response to specific tissue affecting method in form of a remote ischemic preconditioning and will allow to determine the role of sAPPα and BDNF trophic factors and changes in iron metabolism in this process, taking into account the role of hepcidin and vitamin D. Moreover, the present project may contribute to the determination of the role of presented procedures on cells proliferation, as example of anty-tumor proprieties.

Therefore, the results of this project could be a significant step in expanding understanding of the role of ischemic preconditioning in the healthy population (in modulating post-exercise muscle damage, cells proliferation, inflammation process) and the role of iron metabolism and vitamin D in those changes In addition, the knowledge on the protective effect of RIPC procedures and their relation to sAPPα, BDNF changes and protein kinase activity will give overview of its novel activity and use.

Research project objectives

The project aims to:

1. Demonstration whether remote ischemic preconditioning (RIPC) will affect the BDNF, hepcidin and cfDNA concentration;
2. Indicate of whether and how long single RIPC session will affect sAPPα, BDNF and hepcidin concentration, and whether these changes will be accompanied by greater resistance of skeletal muscles to damage induced by eccentric exercises;
3. Show whether training based on a 10-day remote ischemic preconditioning will induce a higher changes of sAPPα, BDNF, hepcidin erytropheron (ERFE) and erythropoietin (EPO) concentration (compared to a single RIPC session);
4. Indicate whether circulating free DNA (cfDNA) may be used as a new early-stage biomarker of muscle damage and training overload durin anaerobic activity.
5. Indicate whether single and 10-day remote ischemic preconditioning training affects vitamin D metabolites concentration changes, and if those changes are Iron dependent.
6. Demonstrate of whether vitamin D binding protein concentration (Gc-Globulin) changes under influence of single and 10-day remote ischemic preconditioning procedures and how it effects vit D metabolites concentration.
7. Show how RIPC and physical activity procedures effects human serum anti-tumor potential, and is it associated with Vitamin D status and Iron metabolism

Hypotheses:

In the project on the basis of current knowledge, the following hypotheses are stated:

1. Remote ischemic preconditioning (RIPC) will increase the concentration of sAPPα and BDNF, which will correlate with higher skeletal muscle resistance to damage;
2. RIPC training will increase the concentration of sAPPα and BDNF, which will persist over a longer period compering to a single RIPC session;
3. Physical activity effects on vitamin D binding protein, megalin, cubilin concentration changes.
4. RIPC procedures and high vit D status protects muscles and reduces oxidative stress induced by physical exercise and protects against oxidative stress induced by high Iron concentration (lower inflammation process and cfDNA concentration).
5. RIPC procedures effects human serum anti-tumor potential against human LNCaP prostate cancer cells.

WORK PLAN

In order to achieve the objectives of the study 60 people will be recruited, then randomly divided into two groups:

* EXPERIMENTAL - REMOTE ISCHEMIC PRECONDICTIONING GROUP (RIPC),
* CONTROL GROUP (C). Furthermore, groups will be divided into subgroups to implement the assumptions of one-time and 10-times RIPC impact on the level of a induced muscle damage and the level of maximum anaerobic capacity. The whole study will be carried out using the assumptions of the experiment - a blank test, and in accordance with the principles of the cross-fertilization experiment.

Experiment Plan:

1. Enrolment of the participants - All untrained subjects will be selected on the basis of the intent letter.
2. Laboratory measurements

   1. anaerobic test (Wingate Anaerobic Test), RIPC 1 time, RIPC 10 times, anaerobic test (Wingate Anaerobic Test),
   2. aerobic test (Bruce Protocol), RIPC 1 time, RIPC 10 times, aerobic test (Bruce Protocol),
   3. evaluation of human serum (from one-time, ten-day RIPC training and placebo populations ) anti-tumor potential on human LNCaP prostate cancer cells
   4. Blood chemistry and molecular analysis
3. Analysis and interpretation of results, preparation of scientific publications
4. Preparation of scientific publications, project settlement

Material The study will be used purposeful selection according to the study inclusion criteria.

4.2 Procedures

The study will consist of six parts:

1. assessment of general health (medical examination), and familiarization with detailed study protocol;
2. assessment of the maximum anaerobic capacity (WAnT);
3. evaluation of one-time and ten-day RIPC training on the level of maximum anaerobic capacity;
4. evaluation of the impact of one-time PostC procedure after WAnT testing, on the level of inflammatory response markers, iron homeostasis, vit D metabolites and BDNF, sAPP α secretion in research groups after 24h rest from WAnT testing;
5. evaluation of human serum (from one-time, ten-day RIPC training and placebo populations) anti-tumor potential on human LNCaP prostate cancer cells;
6. evaluation of selected laboratory exponents in serum and plasma samples collected during the study 24 hours, 48 hours, 72 hours and 120 hours from an episode of muscle damage induced by eccentric exercises;

Each participant will be at hydrated state and before their first meal in the morning hours (8:00-9:00 a.m.). Before proper measures, each participants had one week earlier a familiarisation session with all procedures.

The ischemic procedure will be carried out before the start of the WAnT and eccentric exercises procedures and muscle damage in accordance with the detailed description of the RIPC procedure. Four-fold filling of the flotation flange will be performed by 5 minutes to the value of 200 mm Hg with 5 minutes' rest interval near the attachment of the initial straight thigh muscle. All performed procedures will be carried out under the Doppler USG control to perform full arterial blood flow restriction.

4.4 Measurement of anaerobic power of the lower limbs (Wingate Anaerobic Test) For anaerobic power of the lower limbs measurement Wingate anaerobic test (WAnT) will be conducted on a cycle ergometer (Monark 894E, Peak Bike from Sweden). For each participant, the saddle height will be individually adjusted so that the after the downward stroke knee angle is approximately 170-175°. Before any experimental testing, each individual will perform a 5 min warm-up on the cycle ergometer with tempo of 60 rpm and 1W/kg. After five minutes break, each participant will be asked to pedal with maximum effort for a period of 30 s against a fixed resistive load of 75 g/kg of total body mass. Each participant was instructed to cycle as fast as possible and was given a 3s countdown before the set resistance was applied Verbal encouragement will be given to all participants to maintain their highest possible cadence throughout WAnT. Data from the cyclo ergometer will be recorded via computer with the MCE 5.1 software.

Variables will be analysed as absolute values (W) and relative to body mass (W/kg).

4.5 Blood samples collection and measurements

The methodology of blood collection for diagnostic tests will be strictly dependent on the requirements of a particular designation and comply with the research procedures (established on the basis of literature data). For laboratory analysis, peripheral blood will be collected. in accordance with the plan:

• for WAnT: for one time and 10-day RIPC - before physical exercise (in the early morning, without a meal), immediately after completion of the Wingate test (up to 5 minutes after the test), after 30 minutes of rest period after completion of the Wingate test (30-35 minutes after the test), 60 minutes after, 6h after, 24 hours after WAnT

The intake will be performed in appropriate standardised tubes by qualified medical personnel:

Serum and plasma will be separated from the samples. The general assessment of the homoeostasis state will be based on preliminary laboratory tests. For the qualitative detection of single proteins involved in antioxidant defence western blotting technique will be performed.

For cfDNA analysis: blood will be collected into cell-free DNA tubes before physical exercise (in the morning, on an empty stomach), immediately after the end of trial, 5 minutes and 60 minutes after the end of exercise. Collected material will be stored in a refrigerator or on ice for cfDNA isolation.

cfDNA will be collected into cell-free DNA tubes and isolated using Quick-cfDNA Serum & Plasma Kit according to the manufacturer's protocol. Obtained material will be aliquoted, stored in -200C and subsequently used for further analyses.

All proposed immunoenzymatic procedures will be carried out using available and standardized methods. Most will be designated by the immunoenzyme method (ELISA) or Luminex Systems multiplexing unit. The ELISA test is used to detect specific proteins in the test material using mono or polyclonal conjugated enzyme antibodies. Ready-made reagent ELISA kits will be used. The concentration of the final product will be assessed by measuring the absorption and comparing with the standard solution. The readings will be made on the Elisa Thermo Scientific microplate reader and MAGPIX xPONENT 4.2 System, RUO.

Vitamin D metabolites concentration will be performed using liquid chromatography coupled with tandem mass spectrometry (QTRAP®4500 (Sciex)SH coupled with ExionLC HPLC system). Serum samples will be analysed in the positive ion mode, using electrospray ionisation. The raw data will be collected using LabSolutions LCGC. To process and quantify the collected data, LabSolutions LCGC will be also used. The following Vit. D metabolites will be determined: 25(OH)D3, 24,25(OH)2D3, 3-epi-25(OH)D3, and 25(OH)D2 levels; and the ratios of 25(OH)D3 to 24,25(OH)2D3, and 25(OH)D3 to 3-epi-25(OH)D3.

In order to determine the sAPPα concentration, it will be necessary to completely remove albumin from human plasma. Initial preliminary tests revealed that the linearity and sensitivity of this ELISA is suboptimal due to non-specific binding attributed to the high protein content of unmodified human plasma. Therefore, all plasma samples have to be HSA-immunosubtracted prior to analysis. sAPPα ELISA levels have to be then normalized to total sAPP Western signals (relative units). Procedure involves serum pre-fraction by depleting human serum albumin using human ProteomeLab IgY albumin based on an HSA spinel column (Phenomenex, Torrance, CA). The procedure will be confirmed by preliminary application of the Western Blot method to determine the protein content in the samples subjected to purification. SAPPα levels will be determined using the ELISA method - Immunobiological Laboratories, Gum, Japan.

For protein qualitative detection western blotting technique will be performed. Sample will undergo protein denaturation, followed by gel electrophoresis. A synthetic or antibody (primary antibody) recognises and binds to a specific target protein.

The electrophoresis membrane is washed in a solution containing the primary antibody, before excess antibody is washed off. A secondary antibody is added which recognises and binds to the primary antibody. The secondary antibody is visualised through various methods such as staining, immunofluorescence, and radioactivity, allowing indirect detection of the specific target protein.

4.6. Cytotoxic activity Cell lines and culture conditions. The LNCaP cell line will be cultured in RPMI 1640 medium (Gibco; Rockville, MD, USA) supplemented with 10% fetal bovine serum (FBS) (CULTILAB, Brazil), 100 U/mL of penicillin, and 100 μg/mL of streptomycin, and it was incubated in a humidified atmosphere at 37°C and 5% CO2. The cytotoxic activity will be evaluated: cells were plated onto 96-well microplates (105 cells/mL) in RPMI 1640 supplemented with 10% FBS in the absence or presence of the EEHS (25-200 μg/mL) for 24 h in a humidified atmosphere at 37°C and 5% CO2. After this period, the cells were washed with PBS and resuspended in buffer (0.01 M HEPES, pH = 7.4, 0.14 M NaCl and 2.5 mM CaCl2). The stained cells will be fluorescently labeled and analyzed using an Accuri C6 flow cytometer and specific software.

4.7 Statistical analysis The results will be analysed statistically using Statistica software. Statistical significance will be determined for p < 0.05. The project analyses significance of differences in results, WAnT and laboratory parameters between groups; Significance of changes after WAnT and regression analysis of test results.

Depending on the normal distribution (Shapiro-Wilk test) of the variables and meeting the criteria of homogeneity of variances (Levene's test) the parametric or non-parametric test will be performed. To evaluate the statistical test for the fold-changes of the biochemical markers, it will be log2 transformed.

ELIGIBILITY:
Inclusion Criteria:

* Dependent on the studied population:

  1. Population of not training grope age and morphologically appropriate participation will take part. Participants will be recruited basing on a voluntary letter of intent. All representatives of the analyzed group participating in the pre-qualification research will fill in the physical activity sheet - Global Health Activity Questionnaire - World Health Organization in Polish adaptation. This will allow to eliminate people who report high levels of physical activity (similar to the level of sport training individuals).
  2. Aerobic sport training Population (long distance runners, marathon runners and other). Participants will be recruited basing on a voluntary letter of intent. All representatives of the analysed group participating in the pre-qualification research will fill in the physical activity sheet - Global Health Activity Questionnaire - World Health Organization in Polish adaptation. All participants have to declare minimum 5 marathon run history (similar to the level of sport results during the run).

Exclusion Criteria:

* taking medicines during the study,
* history of cardiovascular disorders,
* history of autonomic nervous system disorders,
* history of mental disorders,
* history of cerebro-cranial traumas,
* history of other diseases that may directly affect obtained results,
* concurrent injuries,
* drugs intake,
* supplements consumption

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 250 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Measurement of the inflammation blood markers using Magnetic Luminex Performance Assays | Change from baseline at 24 hours after fatigue-induced exercise (before and after IPC protocol)
  The intake will be performed in appropriate standardized BD Vacutainer tubes by qualified medical personnel:
  Serum and plasma will be separated from the samples, Each sample to obtain the serum will be centrifuged at 2500-3000 rpm for 10 minutes in 4° C and stored in 1.5 ml tubes at - 80° C until the assay (no longer than 6 months).
  The following secretory factors and markers of inflammation will be determined in serum or blood plasma (depending on the requirements of the method used) and then analysed in detail using immu:
  * high sensitive C-protein (hsCRP),
  * creatine kinas (CK),
  * lactic acid (LA),
  * interleukin 6 (IL6),
  * interleukin 10 (IL10),
  * interleukin 15 (IL15),
Measurement of the Iron metabolism blood markers using Magnetic Luminex Performance Assays and ELISA Assays | Change from baseline at 24 hours after fatigue-induced exercise (before and after IPC protocol)
  The intake will be performed in appropriate standardized BD Vacutainer tubes by qualified medical personnel: Serum and plasma will be separated from the samples, Each sample to obtain the serum will be centrifuged at 2500-3000 rpm for 10 minutes in 4° C and stored in 1.5 ml tubes at - 80° C until the assay (no longer than 6 months). The following secretory factors and markers will be messured:
  * free Iron
  * hepcidin,
  * transferrin,
  * ferritin,
  * EPO,
  * EFRE,
  * TIBC,
Measurement of neurotrophic, angiogenic blood markers using Automated Hematology Analyzers and Magnetic Luminex Performance Assays | Change from baseline at 24 hours after fatigue-induced exercise (before and after IPC protocol)
  The intake will be performed in appropriate standardized BD Vacutainer tubes by qualified medical personnel: Serum and plasma will be separated from the samples, Each sample to obtain the serum will be centrifuged at 2500-3000 rpm for 10 minutes in 4° C and stored in 1.5 ml tubes at - 80° C until the assay (no longer than 6 months). The following secretory factors and markers of inflammation will be determined: angiogenin (ANG), • insulin-like growth factor-1 (IGF-1), • Growth Differentiation Factor 15 (GDF15), • nerve growth factor (NGF), • Amyloid Precursor Protein- α (sAPPα), • angiopoietin (ANGP1), • brain-derived neurotrophic factor (BDNF) • growth differentiation factor 15 (GDF-15), • tumor necrosis factor α (TNFα).
The general assessment of the homoeostasis Automated Hematology Analyzers | Before all procedures and before post-IPC testing
  * blood morphology,
  * glycemia,
  * free iron,
  * activity of alanine aminotransferase (ALT),
  * aspartate aminotransferase (AST),
  * creatine kinase (CK),
  * lactate dehydrogenase (LDH),
  * concentration of insulin,
  * total cholesterole
  * creatinine,

SECONDARY OUTCOMES:
Measurement of proteins involved in antioxidant defence using Western Blotting Techniques | Change from baseline at 24 hours after fatigue-induced exercise (before and after IPC protocol)
  Qualitative detection of single proteins involved in antioxidant defence using western blotting technique. Proteins involved in antioxidant defence, and inflammation will be identified and measured:
  * involved in antioxidant defense (superoxide dismutase [SOD1], SOD2, glutathione peroxidase [GPx]),
  * inflammation (interleukin-6.
Measurement of anaerobic power of the lower limbs (Wingate Anaerobic Test) | Before and after 1-time and 10-times IPC/SHAM procedures
  For anaerobic power of the lower limbs measurement Wingate anaerobic test (WAnT) will be conducted on a cycle ergometer. Data from the cyclo ergometer will be recorded via computer with the MCE 5.1 software.
  The following WAnT variables will be considered:
  * total work value (Wtot),
  * maximum anaerobic power (PPWAnT),
  * maximum power (TUZ),
  * maximum power maintenance (TUT) to 0.01s,
  * power drop (WSM) (%). Variables will be analysed as absolute values (W) and relative to body mass (W/kg).
Messurment of cfDNA changes | Before, and 5 min, 60 min after every WAnT performance
  cfDNA will be collected into cell-free DNA tubes (Roche) and isolated using Quick-cfDNA Serum & Plasma Kit (Zymo Research) according to the manufacturer's protocol. Obtained material will be aliquoted, stored in -200C and subsequently used for further analyses. Blood samples will be collected into cell-free DNA tubes before physical exercise (in the morning, on an empty stomach), immediately after the end of trial, 5 minutes and 60 minutes after the end of exercise. Collected material will be stored in a refrigerator or on ice for cfDNA isolation
Measurement of isolated serum cytotoxic activity | Up to 3 months post-experimental period
  The LNCaP cell line will be cultured in RPMI 1640 medium supplemented with 10% fetal bovine serum (FBS), 100 U/mL of penicillin, and 100 μg/mL of streptomycin, and incubated in a humidified atmosphere at 37°C and 5% CO2. The cytotoxic activity will be evaluated using the method described by Paredes-Gamero with some modifications. Cells will be plated onto 96-well microplates (105 cells/mL) in RPMI 1640 supplemented with 10% FBS in the absence or presence of the EEHS (25-200 μg/mL) for 24 h in a humidified atmosphere at 37°C and 5% CO2. After this period, the cells will be washed with PBS and resuspended in buffer (0.01 M HEPES, pH = 7.4, 0.14 M NaCl and 2.5 mM CaCl2). The stained cells will be fluorescently labeled and analyzed using an Accuri C6 flow cytometer and Accuri C6 software.
Body composition analyses using bioelectrical impedance analysis (BIA) | During the initial visit, and before and after every experimental phase (1-time; 10-times IPC procedures)
  The participant's body mass and height, leg lean mass (LLM) of lower limbs will be measured by a multi-frequency bioelectrical impedance method using the body composition analyser - Inbody 720 (Biospace, Korea, Seoul). Weight and height will be combined to report BMI in kg/m^2, and all specific analyses will give percent of muscle mass in every limb and part of body. The measured values will be served for normalisation of the peak torque outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Jędrzej Antosiewicz, Full Profesor, Principal Investigator — Medical University of Gdańsk, Department of Bioenergetics and Physiology of Exercise, Gdańsk, Poland
Locations (2):
- Poland (2):
  - Gdansk University of Physical Education and Sport, Gdansk, Pomeranian Voivodeship
  - University of Physical Education and Sport (GUPES), Gdansk, Pomeranian Voivodeship

IPD SHARING:
Plan to Share IPD: No
Individual participant data will be shared only on rational wishes from the main researchers

REFERENCES:
- [Background] Paredes-Gamero EJ, Martins MN, Cappabianco FA, Ide JS, Miranda A. Characterization of dual effects induced by antimicrobial peptides: regulated cell death or membrane disruption. Biochim Biophys Acta. 2012 Jul;1820(7):1062-72. doi: 10.1016/j.bbagen.2012.02.015. Epub 2012 Mar 7. PMID 22425533
- [Background] Mockett BG, Richter M, Abraham WC, Muller UC. Therapeutic Potential of Secreted Amyloid Precursor Protein APPsalpha. Front Mol Neurosci. 2017 Feb 7;10:30. doi: 10.3389/fnmol.2017.00030. eCollection 2017. PMID 28223920
- [Background] Mieszkowski J, Kochanowicz M, Zychowska M, Kochanowicz A, Grzybkowska A, Anczykowska K, Sawicki P, Borkowska A, Niespodzinski B, Antosiewicz J. Ferritin Genes Overexpression in PBMC and a Rise in Exercise Performance as an Adaptive Response to Ischaemic Preconditioning in Young Men. Biomed Res Int. 2019 Apr 11;2019:9576876. doi: 10.1155/2019/9576876. eCollection 2019. PMID 31111074
- [Background] Loenneke JP, Wilson JM, Balapur A, Thrower AD, Barnes JT, Pujol TJ. Time under tension decreased with blood flow-restricted exercise. Clin Physiol Funct Imaging. 2012 Jul;32(4):268-73. doi: 10.1111/j.1475-097X.2012.01121.x. Epub 2012 Jan 18. PMID 22681603
- [Background] Boppart MD, Asp S, Wojtaszewski JF, Fielding RA, Mohr T, Goodyear LJ. Marathon running transiently increases c-Jun NH2-terminal kinase and p38 activities in human skeletal muscle. J Physiol. 2000 Aug 1;526 Pt 3(Pt 3):663-9. doi: 10.1111/j.1469-7793.2000.00663.x. PMID 10922016
- [Background] Berchtold NC, Kesslak JP, Cotman CW. Hippocampal brain-derived neurotrophic factor gene regulation by exercise and the medial septum. J Neurosci Res. 2002 Jun 1;68(5):511-21. doi: 10.1002/jnr.10256. PMID 12111841
- [Background] Bar-Or O. The Wingate anaerobic test. An update on methodology, reliability and validity. Sports Med. 1987 Nov-Dec;4(6):381-94. doi: 10.2165/00007256-198704060-00001. No abstract available. PMID 3324256
- [Background] Bailey TG, Jones H, Gregson W, Atkinson G, Cable NT, Thijssen DH. Effect of ischemic preconditioning on lactate accumulation and running performance. Med Sci Sports Exerc. 2012 Nov;44(11):2084-9. doi: 10.1249/MSS.0b013e318262cb17. PMID 22843115
- [Background] Arosio P, Elia L, Poli M. Ferritin, cellular iron storage and regulation. IUBMB Life. 2017 Jun;69(6):414-422. doi: 10.1002/iub.1621. Epub 2017 Mar 27. PMID 28349628
- [Background] Tug S, Mehdorn M, Helmig S, Breitbach S, Ehlert T, Simon P. Exploring the Potential of Cell-Free-DNA Measurements After an Exhaustive Cycle-Ergometer Test as a Marker for Performance-Related Parameters. Int J Sports Physiol Perform. 2017 May;12(5):597-604. doi: 10.1123/ijspp.2016-0157. Epub 2016 Sep 6. PMID 27617485
- [Background] Turner PR, O'Connor K, Tate WP, Abraham WC. Roles of amyloid precursor protein and its fragments in regulating neural activity, plasticity and memory. Prog Neurobiol. 2003 May;70(1):1-32. doi: 10.1016/s0301-0082(03)00089-3. PMID 12927332
- [Background] Vasques JF, Heringer PVB, Goncalves RGJ, Campello-Costa P, Serfaty CA, Faria-Melibeu ADC. Monocular denervation of visual nuclei modulates APP processing and sAPPalpha production: A possible role on neural plasticity. Int J Dev Neurosci. 2017 Aug;60:16-25. doi: 10.1016/j.ijdevneu.2017.03.003. Epub 2017 Mar 18. PMID 28323038
- [Background] de Groot PC, Thijssen DH, Sanchez M, Ellenkamp R, Hopman MT. Ischemic preconditioning improves maximal performance in humans. Eur J Appl Physiol. 2010 Jan;108(1):141-6. doi: 10.1007/s00421-009-1195-2. Epub 2009 Sep 18. PMID 19760432
- [Background] Chen YT, Chen WY, Huang XT, Xu YC, Zhang HY. Iron dysregulates APP processing accompanying with sAPPalpha cellular retention and beta-secretase inhibition in rat cortical neurons. Acta Pharmacol Sin. 2018 Feb;39(2):177-183. doi: 10.1038/aps.2017.113. Epub 2017 Aug 24. PMID 28836584
- [Background] Breitbach S, Tug S, Simon P. Circulating cell-free DNA: an up-coming molecular marker in exercise physiology. Sports Med. 2012 Jul 1;42(7):565-86. doi: 10.2165/11631380-000000000-00000. PMID 22694348
- See also: Metadata — https://zenodo.org/records/15878628